CLINICAL TRIAL: NCT02609919
Title: Assessment of Immediate Adverse Reactions in Children Under 2 Years of Age Following Administration of Gadoteric Acid (Gd-DOTA or Dotarem)
Brief Title: Assessment of Immediate Adverse Reactions From Dotarem in Children Under 2 Years of Age
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Shannon G. Farmakis, M.D., Assistant Professor, St. Louis University
Other Study IDs: Dotarem Study; 26250 (Other: Saint Louis University Institutional Review Board)
Record Dates: First submitted 2015-11-12; First posted 2015-11-20 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Adverse Reaction to Drug; Allergic Reaction to Contrast Media
Keywords: study of contrast reaction in children under 2 years of age; safety
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — gadolinium 1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetraacetate; gadoterate meglumine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gadoteric Acid — MRI Contrast Agent
  Other Names: Gd-DOTA; Dotarem

SUMMARY:
Our primary outcome is to assess the safety of Dotarem in children <2 years old up to 24 hours after Dotarem injection. Patients will be monitored for any adverse events that occur for 2 hours following the completion of the MRI exam. The type of event, time of onset, duration of symptoms, intensity of the reaction (mild, moderate, severe), causality (not related, probably related, related, definitely related, unclassifiable), and subsequent outcome (required treatment, favorable outcome, recovery with sequela, or death) will be documented. Parents will be given instruction sheets on who and when to call should any adverse event occur after discharge. Parents will be called by the radiology department the next day to identify any adverse events that occurred during the first 24 hours after discharge from the hospital.

Our secondary outcome is to assess image quality of the exam. The pre-contrast images will be compared to the combined pre- and post-contrast images following administration of Dotarem by radiologists who are blinded to the patients' clinical information to assess for improvement of image quality and delineation of structures with contrast.

DETAILED DESCRIPTION:
Our primary outcome is to assess the safety of Dotarem in these patients up to 24 hours after Dotarem injection. The patients will be monitored in the hospital for at least 2 hours following the completion of the MRI exam. Many of these patients will have received sedation for the MRI and would be monitored normally for up to 1 hour after the exam is completed. Patients will be monitored for any adverse events that occurred during the observation period. The type of event, time of onset, duration of symptoms, intensity of the reaction (mild, moderate, severe), causality (not related, probably related, related, definitely related, unclassifiable), and subsequent outcome (required treatment, favorable outcome, recovery with sequela, or death) will be documented. Parents will be given an information sheet prior to discharge indicating the possible adverse events that may occur related to the administration of Dotarem with instructions on what to do and who to call, if necessary, should any of them occur. Parents will be called by the radiology department the next day to identify any adverse events that occurred during the first 24 hours after discharge from the hospital.

Our secondary outcome is to assess image quality of the exam. The pre-contrast images will be compared to the combined pre- and post-contrast images following administration of Dotarem by radiologists who are blinded to the patients' clinical information to assess for improvement of image quality and delineation of structures with contrast.

200 patients are expected to be enrolled in this study over the course of 18 months.

Exclusion criteria: Patients 2 years of age or older. Patients receiving an MRI exam without contrast. Patients with a GFR <30. Patients with known renal failure or prior gadolinium based contrast agent hypersensitivity reaction. Patients who receive an MRI exam using a different gadolinium-based contrast agent. Patients who are not accompanied by a parent will not be included. Patients who are unable to complete the MRI exam prior to contrast administration will be excluded.

Inclusion criteria: Any patient under 2 years of age undergoing an MRI exam of the neuraxis or body with and without contrast as part of their standard of care. Included patients may be scheduled with simultaneous sedation for the MRI. Nonsedated patients also qualify for the study.

Patients who qualify for Dotarem administration are usually preselected by the radiologist depending on the type of exam and the reason for the study. While, the use of Dotarem is not approved by the FDA in this patient population, off-label use of the agent is routinely performed during routine clinical care of patients in this age group in our practice. Those patients who would be given Dotarem as part of routine standard of care will be asked to enroll. Written consent will be obtained from the parents. Patients will be recruited over an 18 month period of time.

All MRI exams will be performed on our 3T GE Discovery 750W or 1.5T GE Signa HDXT 23.0.

All patients will have the following information recorded: age, sex, weight, risk factors (renal disease, cardiac disease, autoimmune disease, dehydration, other medical conditions), reason for exam, type of exam, dose of Dotarem, route of injection (manual or power injection), a premedication regimen (i.e. steroids), and tolerance to injection. In addition, when applicable, the types of medications used for sedation will be recorded as well as the route of sedation: deep sedation, laryngeal mask airway, or general endotracheal anesthesia.

Patients will be given a weight-based dose of Dotarem of 0.2mL/kg (0.1 mmol/kg) body weight. It will be administered as an intravenous bolus injection at a flow rate of approximately 1-2 mL/second either by manual or power injection.

During the MRI exam, all patients will undergo continuous monitoring of heart rate and peripheral oxygen saturation. Sedated patients will be monitored similarly until they reach an Aldrete score >6. After this the monitoring devices will be removed. The patients will then be observed off the monitors until a total of 2 hours after the exam has elapsed.

All adverse drug events (ADEs) will be documented including nausea, headache, injection site pain, injection site coldness, burning sensation, heart arrhythmia, allergic reactions (cardiac or respiratory arrest, laryngeal edema, angioedema, urticarial, seizures, syncope, tremors, muscle spasms or weakness, diarrhea, drooling, and fever. If an ADE occurs, the timing related to the injection of Dotarem will be recorded.

A crash cart is available directly across the hallway from the MRI suite in the Sedation/Nursing area in radiology. Nursing staff and a staff radiologist are available at all times for immediate reactions. If a severe anaphylactic or bronchospasm reaction occurs, the patient will be brought to the Emergency Department. Management and treatment of acute reactions to contrast media will follow the guidelines outlined in Table 4 of the ACR Manual on Contrast Media Version 10.1 (2015).

Aldrete Scoring System:

Activity Voluntary movement of all limbs to command 2 Voluntary movement of 2 extremities to command 1 Unable to move 0 Respiration Able to breathe deeply and cough 2 Dyspnea, hypoventilation 1 Apnea 0 Circulation B/P + 20% of pre-anesthetic level 2 B/P + 20%-50% of pre-anesthetic level 1 B/P + 50% of pre-anesthetic level 0 Consciousness Fully awake 2 Arousable 1 Unresponsive 0 Color Pink 2 Pale, dusky, blotchy, jaundice, other 1 Cyanotic 0

Phone Call: The follow up phone call to the parents the next day (>24 hours) will include asking the parents the following questions:

Did your child experience any of the following after being discharged from the hospital from the MRI exam? Headache Y/N Nausea Y/N Dizziness Y/N Dysgeusia Y/N Feeling Hot Y/N Injection site reactions Y/N Vomiting Y/N Rash (includes generalize, macular, popular, pruritic) Y/N Erythema Y/N Hypersensitivity/Anaphylactoid (i.e. urticarial, facial edema, eyelid edema, flushing, cough, sneezing, wheezing, chest pain, cyanosis) Y/N Dyspnea Y/N Paresthesia Y/N

Following your child's discharge from MRI, did he/she have any other clinic appointments or tests/exams in the hospital? If so, what were they?

Our secondary outcome is to assess the image quality of the exam. Patients will initially undergo a pre-contrast MRI examination followed by the administration of Dotarem. The pre-contrast images will be compared to the combined pre- and post-contrast images independently by 3 radiologists blinded to the clinical information. The three primary imaging components judged will be contrast enhancement, border delineation, and internal morphology. In addition, within each of these components, the radiologist will assign a result based on a pre-defined scoring scale. These include the following:

Pre-contrast images vs. Paired pre-post contrast images:

Border delineation: better, same, not better, missing Internal morphology: better, same, not better, missing Contrast enhancement: better, same, not better, missing

Better is defined as those patients in which the combined pre- and post-contrast exam images were greater than the pre-contrast images alone. Same is defined as those patients in which the characteristics of a lesion or disease did not change following contrast administration because of the inherent characteristics of the lesion/disease in which enhancement is not expected. Missing identifies those patients in which a score was not assigned.

ELIGIBILITY:
Inclusion Criteria:

* Any patient under 2 years of age undergoing an MRI exam of the neuraxis or body with or without and with contrast as part of their standard of care.
* Included patients may be scheduled with simultaneous sedation for the MRI.
* Nonsedated patients also qualify for the study.

Exclusion Criteria:

* Patients 2 years of age or older.
* Patients receiving an MRI exam without contrast.
* Patients with a GFR <30.
* Patients with known renal failure or prior gadolinium based contrast agent hypersensitivity reaction.
* Patients who receive an MRI exam using a different gadolinium-based contrast agent.
* Patients who are not accompanied by a parent will not be included.
* Patients who are unable to complete the MRI exam prior to contrast administration will be excluded.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under 2 years of age requiring MRI with Contrast
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-01; Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
number and type of adverse drug events following the administration of gadoteric acid (Gd-DOTA or Dotarem) as well as when these reactions occur | 18 months
  Safety and efficacy

SECONDARY OUTCOMES:
Image quality | 18 months
  To assess whether lesion detection and characterization is improved with Dotarem compared to the noncontrast images.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Farmakis, MD, Principal Investigator — St. Louis University School of Medicine
Locations (1):
- Saint Louis University, St Louis, Missouri, United States